CLINICAL TRIAL: NCT04891393
Title: The Effects of Caffeine on Human Spinal Motoneurons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 26014
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Motor Neuron; Excitability; Caffeine
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): Single-dose, orally ingested, instant coffee.
  Interventions: Dietary Supplement: Coffee
- Inactive Placebo (Placebo Comparator): Single-dose, orally ingested, instant decaffeinated coffee (equal weight to intervention dose).
  Interventions: Dietary Supplement: Decaffeinated coffee

INTERVENTIONS:
Dietary Supplement: Coffee — Starbucks brand "Via" instant coffee. (Caffeine Content: 3 mg / kg)
  Arms: Caffeine
Dietary Supplement: Decaffeinated coffee — Starbucks brand "Via" instant decaffeinated coffee. (Caffeine Content: 15 - 25 mg)
  Arms: Inactive Placebo

SUMMARY:
This study evaluates the effects of orally ingested, commercially available, coffee (3 mg/kg of caffeine) on the excitability of human spinal motoneurons of the lower leg.

DETAILED DESCRIPTION:
Recently, it has been shown that human spinal motoneurons do not simply act as a binary control system. Instead, they are regulated by intrinsic properties that can elicit lingering effects on the descending motoneuron. Caffeine, one of the world's most popular over-the-counter supplements, can potentially augment these characteristics of motoneurons. Using decomposition software and non-invasive, high-density surface electromyography, it is possible to extract the characteristics of these motoneurons. This project will utilize a double-blind, inactive-placebo controlled, crossover design study to examine and quantify the effects of caffeine on motoneuron excitability.

ELIGIBILITY:
Inclusion Criteria:

● Between 18 and 70 years of age

Exclusion Criteria:

* Significant neurological or orthopedic injuries, which may limit volitional torque generation in the tested muscles.
* Significant change in the subjects' health or treatment in the past month.
* Known history of cardiovascular pathology (to include: uncontrolled hypertension, cardiac arrhythmias) or medical restrictions to caffeine ingestion.
* Allergies or dislike of coffee.
* Women who are pregnant will be excluded due to potential forces at trunk from pelvic safety harness and due to potential adverse effects of caffeine on the developing child.
* Women who are breastfeeding will be excluded due potential adverse effects on the breastfeeding infant from caffeine administration.
* Adults unable to consent, minors, pregnant women, and prisoners will not be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Motoneuron excitability (Delta-f) | Measured repeatedly at set intervals; Pre-Intervention & 30, 60, 90 minutes post-Intervention
  Changes in motorneuron excitability, as quantified by Delta-F values. A paired motor unit technique will be utilized (Gorassini et al., 2002). (Typically, these values range from -5 to +10).

SECONDARY OUTCOMES:
Motor Unit Discharge Rate | Measured repeatedly at set intervals; Pre-Intervention & 30, 60, 90 minutes post-Intervention
  Changes in motor unit discharge rate. This is a single value that ranges from, approximately, 0 to 30.
Coherence | Measured repeatedly at set intervals; Pre-Intervention & 30, 60, 90 minutes post-Intervention
  Changes in coherence values. Coherence provides a normalized value of the strength of correlation in the frequency domain. The magnitude of the correlation of the Fourier transforms of two spike trains is squared producing a value between 0 and 1, with 1 corresponding to a perfect linear prediction at a particular frequency (Rosenberg et al., 1989). This will be calculated using the composite spike train (Negro & Farina, 2012) and, finally, z-transformed to allow for between-trial comparisons.
Motor Unit Recruitment Threshold | Measured repeatedly at set intervals; Pre-Intervention & 30, 60, 90 minutes post-Intervention
  Changes in motor unit recruitment threshold. As assessed by determining the amount of force (percentage of maximum volitional force output) needed to recruit an individual motor unit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Thompson, PT, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorassini M, Yang JF, Siu M, Bennett DJ. Intrinsic activation of human motoneurons: possible contribution to motor unit excitation. J Neurophysiol. 2002 Apr;87(4):1850-8. doi: 10.1152/jn.00024.2001. PMID 11929906
- [Background] Rosenberg JR, Amjad AM, Breeze P, Brillinger DR, Halliday DM. The Fourier approach to the identification of functional coupling between neuronal spike trains. Prog Biophys Mol Biol. 1989;53(1):1-31. doi: 10.1016/0079-6107(89)90004-7. No abstract available. PMID 2682781
- [Background] Farina D, Negro F. Accessing the neural drive to muscle and translation to neurorehabilitation technologies. IEEE Rev Biomed Eng. 2012;5:3-14. doi: 10.1109/RBME.2012.2183586. PMID 23231985